CLINICAL TRIAL: NCT04240145
Title: Non Alcoholic Steatohepatitis in Relation to Visceral and Subcutaneous Fat
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gehad Abd Elaziz Mhmoud Ahmad (Other)
Responsible Party: Sponsor-Investigator, Gehad Abd Elaziz Mhmoud Ahmad, Assiut Universityhospital, Assiut University
Organization: Assiut University (Other)
Other Study IDs: NASH
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2019-10

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MSCT Abdomen — Visceral fat volumetry using MSCT and it's relation to NASH

SUMMARY:
Evaluate the relationship between the severity of fatty liver in NAFLD assessed by ultrasonography and CT and the visceral fat area measured by CT

DETAILED DESCRIPTION:
Non alcoholic fatty liver disease is one of the most common causes of chronic liver disease world wide . Severe forms of NAFLD such as nonalcoholic steatohepatitis can progress to end-stage liver disease such as cirrhosis or hepatocellular carcinoma. Therefore, investigating risk factors associated with hepatic steatosis is required to perform effective screening .

Hepatic steatosis develops for a variety reasons but obesity is the most common associated condition.

Obesity is considered a gateway disease and NAFLD is considered to be one of the phenotypes of metabolic syndrome, which is characterized by obesity with visceral fat accumulation, diabetes, hypertension and dyslipidemia.

Individuals with severe obesity have a disproportionately high risk of comorbidities including nonalcoholic fatty liver disease (NAFLD), cardiovascular disease and diabetes.

The distribution of fat appears more important than the total fat mass in obesity .A predominantly upper body fat distribution increases the risks for the metabolic complications of obesity including hepatic steatosis especially when it is associated with increased intra abdominal fat .

Most "metabolically obese" normal weight subjects have some increase in adipose tissue mass and insulin resistance probably due to an increase in visceral fat. Thus, subjects with a relatively low BMI can have gross increases in abdominal visceral fat, and others with a high BMI may have very little intra abdominal/visceral fat .

Several studies suggested visceral adiposity to be a clinical predictor of hepatic steatosis .

In addition, the severity of fatty liver has been linked to the VAT area as evaluated by CT.

ELIGIBILITY:
Inclusion Criteria:

* patient aged from 18years to 75years of both gender presented to Alrajhi hospital with raised liver enzymes in period from October 2019 to June 2020

Exclusion Criteria:

* patient with viral hepatitis History of drug intake Auto immune hepatitis

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient from age 18 to 75 years of both gender presented to Assiut University hospital with raised liver enzymes
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
NasH in relation to visceral and subcutaneous fat | base line
  Visceral fat volumetryusing MSCT and it'srelation tovisceral andsubcutaneous fat

CONTACTS AND LOCATIONS:
Overall Officials: Assiut University, Principal Investigator — Assiut University

REFERENCES:
- [Background] Kershaw EE, Flier JS. Adipose tissue as an endocrine organ. J Clin Endocrinol Metab. 2004 Jun;89(6):2548-56. doi: 10.1210/jc.2004-0395. PMID 15181022
- [Background] Angulo P. Nonalcoholic fatty liver disease. N Engl J Med. 2002 Apr 18;346(16):1221-31. doi: 10.1056/NEJMra011775. No abstract available. PMID 11961152
- [Background] Ong JP, Pitts A, Younossi ZM. Increased overall mortality and liver-related mortality in non-alcoholic fatty liver disease. J Hepatol. 2008 Oct;49(4):608-12. doi: 10.1016/j.jhep.2008.06.018. Epub 2008 Jul 9. PMID 18682312